CLINICAL TRIAL: NCT04695782
Title: Pencil Beam Proton Therapy for Pelvic Recurrences in Rectal Cancer Patients Previously Treated With Radiotherapy
Acronym: ReRad II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCPT221020
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neo-adjuvant pencil beam proton therapy: 55 Gy(RBE)/44fx (1.25 Gy per fraction), two daily (Experimental)
  Interventions: Radiation: Pencil beam proton radiotherapy
- Definitive arm pencil beam proton therapy: 57.5-65Gy(RBE)/46-52 fx (1.25 per fraction) two daily (Experimental)
  Interventions: Radiation: Pencil beam proton radiotherapy

INTERVENTIONS:
Radiation: Pencil beam proton radiotherapy — Doseescalated pencil beam proton Therapy

SUMMARY:
Study design:

A prospective phase II, non-randomized observational study of dose-escalated pencil beam proton therapy re-irradiation for pelvic recurrences from rectal cancer.

Re-irradiation is either a part of neo-adjuvant treatment or as a definitive treatment strategy for un-resectable recurrences.

ELIGIBILITY:
Inclusion Criteria:

* • Locally recurrent rectal cancer.

  * Bioptically verified (adenocarcinoma )
  * Available dose plan from primary radiotherapy
  * Previous pelvic RT (>30Gy EQD2)
  * Evaluated in MDT-conferences (Herlev, Aarhus)
  * Age>18 years
  * PS 0-2
  * Adequate organ function
  * Informed consent

Exclusion Criteria:

* Non-resectable distant metastases (PET-CT)
* Unable to undergo MRI, PET-CT
* Inability to attend full course radiotherapy and follow up in the out patient clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
R0-resection | 5-6 years
  Neo-adjuvant treatment: Rate of pathological complete resection (R0)
1-year local control | 6-7 years
  Definitive treatment: Rate of 1-year local control rates evaluated by CT or MRI.

SECONDARY OUTCOMES:
Local recurrence | 6-8 years
  Local re-recurrence determined by imaging 6, 12 and 24 month post treatment
Disease free survival | 10 years
  Disease free survival, defined as time from first day of treatment until first documented sign of disease or death from any course
Overall survival | 10 years
  Overall survival defined as time from first day of treatment to death from any cause
Toxicity | 5-7 years
  Toxicity evaluated by NCI-CTCAE v. 5.0 acute and chronic
Patient reported outcomes | 5-7 year
  Quality of life assessment by EORTC QLQ-c30, QLQ-CR29, supplementary EORTC items, and LARS score. Acute and chronic

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Centre for Particle Therapy, Aarhus, Denmark